CLINICAL TRIAL: NCT02305732
Title: A Prospective, Open Label, Treatment Use Study of Patient Safety Following Transfusion of INTERCEPT Platelet Components
Acronym: TRUE
Status: Completed | Type: Observational
Sponsor: Cerus Corporation (Industry)
Collaborators: American National Red Cross (Other)
Responsible Party: Sponsor
Other Study IDs: CLI 00108
Record Dates: First submitted 2014-11-25; First posted 2014-12-03 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2017-12

CONDITIONS: Chikungunya Virus; Dengue Virus
Keywords: Chikungunya virus; CHIKV; Dengue virus; DENV; pathogen inactivation; platelets; Puerto Rico

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Biological: INTERCEPT Platelets — INTERCEPT platelet components (PC). Leukocyte reduced apheresis platelet components collected in Platelet Additive Solution (PAS) or 100% plasma without gamma irradiation, bacterial detection, and Cytomegalovirus (CMV) serology testing.

SUMMARY:
The rationale for a Treatment Use Investigational Device Exemption (IDE) of INTERCEPT PCs is to address current gaps in platelet transfusion safety in selected geographic regions. The objective is to provide access to INTERCEPT PCs for patients who might be at risk of transfusion-transmitted infection (TTI) due to Chikungunya virus (CHIKV) and Dengue virus (DENV) in regions in which a substantial proportion of the population has been infected or is at risk of infection by these pathogens (Petersen 2014); and the risk of asymptomatic infection among qualified blood donors is recognized (Stramer 2012, Adda 2014).

The study is designed as a prospective, open label, multi-center, observational study to evaluate the safety and efficacy of INTERCEPT platelet components.

DETAILED DESCRIPTION:
Upon written informed consent, patients will be transfused with study PCs according to local practices. Each patient will be supported with platelets as clinically indicated in a manner that is consistent with the local standard of care. The study will be conducted in two phases. During the pilot phase, patients will sign informed consent to have study data collected following transfusion with conventional PCs. The objective of the pilot phase is to evaluate study logistics and data collection methods. During the INTERCEPT Treatment Use phase, patients will sign informed consent to receive INTERCEPT PCs, provide blood samples, and collect study data (demographics, transfusion data, and safety data).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a serious disease expected to require or requiring a transfusion of platelet component(s)
* Patient population as defined by each Investigator and their institutional review board (IRB).
* Patient provides written informed consent

Exclusion Criteria

* Documented allergy to psoralens
* Neonatal patients treated with phototherapy devices that emit wavelengths less than 425 nm due to the potential for erythema resulting from interaction between ultraviolet light and amotosalen.
* Pregnant women in their third trimester of pregnancy (due to possibility the neonate may need bilirubin light treatment after birth).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring a platelet transfusion.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Stramer, PhD, Principal Investigator — American National Red Cross
Locations (8):
- Puerto Rico (8):
  - Hospital General Menonita de Aibonito, Aibonito
  - Hospital General Menonita de Caguas, Caguas
  - Hospital General Menonita de Cayey, Cayey
  - Center Hospital Manati, Manatí
  - Hospital San Lucas Ponce, Ponce
  - Hospital La Concepcion San German, San Germán
  - Centro Cardiovascular de Puerto Rico and the Caribbean, San Juan
  - Veteran Administration, San Juan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- INTERCEPT: Includes patients enrolled during the INTERCEPT-Treatment-Use phase of the study who received at least one INTERCEPT platelet component.
Period: Overall Study
Arm/Group | INTERCEPT
Started | 90
Completed | 72
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | INTERCEPT
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 50
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 90

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Transfused INTERCEPT Platelet Components With a Post-treatment Platelet Dose ≥ 3.0×10^11 Platelets.
Description: INTERCEPT platelet components (PCs) manufactured for this study are leukocyte reduced apheresis PCs processed using the INTERCEPT Blood System (IBS) for platelets. The IBS for platelets is a Class III medical device approved by the FDA for the ex-vivo preparation and storage of pathogen reduced apheresis PCs. The system is used to inactivate a broad range of pathogens, including viruses, bacteria, and protozoan parasites as well as contaminating donor leukocytes. Post-manufacturing, INTERCEPT PCs are either transfused or stored according to blood center standard operating procedures, US FDA, and AABB Guidelines.
  Subjects enrolled in this study are transfused with INTERCEPT PCs as dictated by the treating physician. One platelet component was treated as one platelet transfusion for the purpose of data analysis in this study.
Time Frame: 1 year
Population: This outcome summarizes the 256 INTERCEPT platelet components transfused during the INTERCEPT-Treatment-Use phase of the study. A total of 90 patients received at least one INTERCEPT platelet component. "1 Transfusion = 1 Intercept Platelet Component".
Measure: Count of Units; unit: Platelet Components
Units Other Than Participants: Platelet Components
Groups:
- Transfused INTERCEPT Components: Includes all INTERCEPT platelet components transfused during the INTERCEPT-Treatment-Use phase of the study.
Arm/Group | Transfused INTERCEPT Components
Number analyzed (Participants) | 90
Number analyzed (Platelet Components) | 256
Platelet Components | 256

2. Primary Outcome: The Proportion of Patients With a Confirmed Case of Transfusion-transmitted Chikungunya Virus or Dengue Infection
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT
Number analyzed (Participants) | 90
Participants | 0

3. Primary Outcome: The Proportion of Patients With Any Transfusion Reactions
Description: Transfusion reactions are defined as adverse events assessed as possibly, likely/probably or certainly related to the INTERCEPT platelet component transfused.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT
Number analyzed (Participants) | 90
Participants | 3

4. Primary Outcome: The Proportion of Patients With Any Unrelated Adverse Event
Description: Unrelated adverse events are defined as adverse events unrelated to the INTERCEPT platelet component transfused.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT
Number analyzed (Participants) | 90
Participants | 26

5. Primary Outcome: The Proportion of Transfused INTERCEPT Platelet Components Associated With Any Transfusion Reactions and/or Unrelated Adverse Event
Description: Transfusion reactions are defined as adverse events assessed as possibly, likely/probably or certainly related to the INTERCEPT platelet component transfused.
  Unrelated adverse events are defined as adverse events unrelated to the INTERCEPT platelet component transfused.
  ""1 Transfusion = 1 Intercept Platelet Component".
Time Frame: 1 year
Population: This outcome summarizes the 256 INTERCEPT platelet components transfused during the INTERCEPT-Treatment-Use phase of the study. A total of 90 patients received at least one INTERCEPT platelet component.
Measure: Count of Units; unit: Platelet Components
Units Other Than Participants: Platelet Components
Arm/Group | Transfused INTERCEPT Components
Number analyzed (Participants) | 90
Number analyzed (Platelet Components) | 256
Platelet Components | 50

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 24 hours following each study transfusion and serious adverse event data were collected for 7 days post each study transfusion.
Arm/Group | INTERCEPT
All-Cause Mortality (participants affected / at risk) | 17/90
Serious Adverse Events (participants affected / at risk) | 19/90
Other Adverse Events (participants affected / at risk) | 15/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTERCEPT (N=90)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 6 (6)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vena cava thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTERCEPT (N=90)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Blood pressure decreased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
HIV test positive (Investigations) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No